CLINICAL TRIAL: NCT07115173
Title: A Single-Center, Single-Arm Clinical Trial to Evaluate the Efficacy of Probit-Based Triple Therapy for Helicobacter Pylori Eradication
Brief Title: Clinical Trial to Evaluate the Efficacy of Probit-Based Triple Therapy for Helicobacter Pylori Eradication
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAQBO_IIT_H.pylori
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Helicobacter Infection
MeSH Terms: conditions — Helicobacter Infections | interventions — Clarithromycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This study aims to evaluate the efficacy and safety of a 14-day triple therapy regimen consisting of (Experimental)
  Interventions: Drug: This study aims to evaluate the efficacy and safety of a 14-day triple therapy regimen consisting of Zastaprazan 20 mg, clarithromycin, and amoxicillin for the eradication of Helicobacter pylori.

INTERVENTIONS:
Drug: This study aims to evaluate the efficacy and safety of a 14-day triple therapy regimen consisting of Zastaprazan 20 mg, clarithromycin, and amoxicillin for the eradication of Helicobacter pylori. — This study aims to evaluate the efficacy and safety of a 14-day triple therapy regimen consisting of Zastaprazan 20 mg, clarithromycin, and amoxicillin for the eradication of Helicobacter pylori.

SUMMARY:
This is a single-center, open-label, non-randomized, single-arm clinical study. Eligible participants who provide written informed consent will undergo screening based on inclusion/exclusion criteria. Enrolled subjects will receive the investigational treatment: Zastaprazan 20 mg (twice daily), clarithromycin 500 mg (twice daily), and amoxicillin 1000 mg (three times daily) for 14 days. Four to eight weeks after completing the therapy, participants will return for a urea breath test to assess H. pylori eradication. The study will also investigate the efficacy of this therapy in clarithromycin-resistant patients to indirectly assess the potential of a dual regimen using Zastaprazan and amoxicillin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 19 to 75 years at consent.
2. Confirmed H. pylori positive by urease breath or enzyme test.
3. Require eradication therapy due to at least one condition: chronic atrophic gastritis, peptic ulcer, history of early gastric cancer or adenoma resection, functional dyspepsia, low-grade MALT lymphoma, idiopathic thrombocytopenic purpura, iron deficiency anemia, hyperplastic polyps, or family history of gastric cancer.
4. Agree to use medically acceptable contraception during the trial (including medically sterile women such as menopausal, hysterectomy, tubal ligation, or bilateral oophorectomy).
5. Provide voluntary written informed consent.

Exclusion Criteria:

1. History of receiving H. pylori eradication therapy prior to study participation.
2. Known hypersensitivity to the investigational product, penicillin-class antibiotics, or macrolide-class antibiotics.
3. Current use of medications contraindicated with the investigational product or concomitant therapy.
4. Abnormal laboratory values in blood chemistry tests as defined by the protocol.
5. pregnant or nursing women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 4 to 8 weeks
  Efficacy of H. pylori eradication therapy. confirmed by negative UBT test

IPD SHARING:
Plan to Share IPD: Undecided